CLINICAL TRIAL: NCT03848858
Title: The Efficacy of Eye Movement Desensitization and Reprocessing Therapy Versus Treatment-As-Usual in a Pilot Randomized Controlled Trial in Reducing Clinical Symptoms and Biological Markers of HIV in Patients With a Recent Diagnosis of HIV
Brief Title: Efficacy of EMDR Therapy, as Compared to Treatment as Usual, in Reducing Clinical Symptoms in People With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: EMDR Europe (Industry); Fundacion IMIM (Other)
Responsible Party: Principal Investigator, Ana Moreno Alcázar, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/8199/I
Record Dates: First submitted 2018-11-07; First posted 2019-02-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS; Psychological Trauma; PTSD
Keywords: HIV; Psychological Trauma; Eye Movement Desensitization and Reprocessing Therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Psychological Trauma; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from the Infectious Diseases Unit of the Hospital del Mar, Barcelona, Spain, and evaluations and therapy sessions will be carried in the Hospital del Mar and in the Hospital del Mar Research Institute. The study consists of a single-blind RCT with two parallel branches, 1) individual therapy with EMDR and TAU, and 2) TAU only, with participants matched by age, sex, and prior trauma burden. Following the initial evaluation, participants will be randomized to either receive up to 6 months of weekly 1 hour EMDR sessions (20 sessions) in addition to the standard medical treatment, or standard medical treatment only. The participants will be evaluated pre- and post- treatment.
Who Masked: Outcomes Assessor
Masking Description: Evaluators will be blind to treatment. Participants cannot be blind to treatment due to the impossibility of creating a sham alternative to EMDR therapy, due to its use of bilateral stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR plus TAU (Experimental): 20 individual weekly sessions of 60 minutes each of Eye Movement Desensitization and Reprocessing Therapy (EMDR), plus Treatment as Usual (TAU), applying first the standard EMDR protocol (Shapiro, 2005), and then a specific protocol for the sequelae of somatic illness and medical trauma (Hase, 2018).
  Interventions: Behavioral: EMDR plus TAU
- TAU only (No Intervention): The patients in this condition are newly diagnosed and will be introduced to the study in their first appointment with the Infectious Diseases Unit, in which analyses of HIV-related biological markers are taken. In a follow up appointment between 1 and 2 weeks later, antiretroviral treatment is initiated. There is a further check-up 1-2 months after initiating antiretroviral treatment, and then 6-monthly check-ups. In these checkups, measures of CD4 and the CD4/CD8 ratio are taken and treatment adherence is reviewed. The patients receiving EMDR therapy will also participate in these activities.

INTERVENTIONS:
Behavioral: EMDR plus TAU — The standard EMDR protocol will first be applied, consisting of 8 phases: 1) Patient history; 2) Patient preparation; 3) Evaluation of the main aspects of the traumatic memory; 4) Desensitization of the memory; 5) Installation of the positive cognition; 6) Body scan; 7) Close and 8) Reevaluation. The specific protocol for the sequelae of somatic illness and medical trauma is next applied. It first focuses on processing past memories related to diagnosis, symptom development, medical procedures and unjust or stressful behaviour with the medical system. Once these are processed, the intervention addresses current symptoms, impairments and triggers. Finally, the patient is helped to face the future and reduce avoidance of medical procedures, avoidance of social life and fear of dying.
  Arms: EMDR plus TAU

SUMMARY:
People living with HIV may suffer HIV-related psychological trauma. Studies also show that this group is vulnerable to non-HIV-related trauma. Trauma can increase vulnerability to stress and reducing the ability to cope. It can have a negative impact on treatment adherence, treatment outcomes, functioning and health-related quality of life. However, despite evidence showing psychological trauma can contribute to poor outcomes in HIV, little research has been carried out to assess whether psychological trauma-focused therapy can help people living with HIV.

A first-line treatment for psychological trauma is Eye Movement Desensitization and Reprocessing (EMDR) therapy. This therapy is recommended by the World Health Organization for treating Post-Traumatic Stress Disorder, with many studies showing this treatment is safe and effective for this disorder. However, it has not to our knowledge been specifically tested in the population of people living with HIV. This project will test whether EMDR therapy, in addition to the standard medical treatment received at the Infectious Diseases Unit, is more effective than standard medical treatment alone in reducing psychological trauma, improving health-related quality of life and improving HIV outcomes in people recently diagnosed with HIV. To test this, the investigators will recruit 40 people who have received a diagnosis of HIV within the last month. 20 will be offered the possibility to receive EMDR treatment for one hour weekly for up to 6 months, in addition to the standard medical treatment, while the other 20 will be offered only the standard medical treatment. The hypotheses of the present study are that the participants who receive EMDR therapy on top of their standard medical treatment will show a reduction in psychological trauma and related symptoms such as anxiety, depression and global distress, as compared to those who did not. The investigators also predict that the EMDR group will show improved functioning and health-related quality of life. The final hypotheses are that the EMDR group will show improved treatment adherence and HIV outcomes. If this study shows that a psychological trauma-focused therapy can help people adjust to a recent HIV diagnosis and have better outcomes, this will have important implications for improving care for people living with HIV.

DETAILED DESCRIPTION:
Background

The seropositive population are vulnerable to high rates of psychological trauma with 30-40% of people living with HIV having HIV-related trauma, and rates of up to 90% of trauma unrelated to HIV. HIV-related trauma is linked to various events such as receiving the diagnosis, the number of medical symptoms, receiving treatment, the level of perceived stigma related to HIV, and witnessing HIV-related deaths. The risk of suffering trauma related to HIV is higher in those with prior trauma and negative life event.

Trauma is known to not only have a serious impact on mental health, but also to be a key predictor of poor prognosis in HIV, affecting treatment outcomes and health-related quality of life. Trauma exposure and the development of trauma symptoms impair psychosocial functioning, increase vulnerability to stress and burden the physiological systems involved in coping and adaptation. Patients with posttraumatic symptoms show poorer treatment adherence, yet even in therapy-adherent individuals, posttraumatic symptoms are associated with immune dysregulation, leading to decreased CD4 cell count and thus negative health outcomes. Trauma-affected patients are also more likely to engage in risky health-related behaviors and to suffer higher functional impairment not explained by CD4 count variance.

Due to the negative impact of trauma in terms of psychological distress and poorer HIV outcomes, psychological interventions which specifically address trauma are needed as an adjunct to antiretroviral treatment, in order to reduce unnecessary mortality related to poor treatment adherence and to improve health-related quality of life and functionality. There is even potential for psychological interventions to impact directly on HIV disease progression. Limited evidence suggests that psychological interventions targeting trauma can have a positive impact on HIV symptom experience, while a small but promising body of research into Mindfulness-based interventions targeted at reducing stress show they may have a positive impact on the biological HIV marker CD4. Therefore, a brief yet effective psychological intervention at the point of diagnosis could have a significant impact in reducing psychological trauma and distress and improving treatment adherence and thus prognosis, and may even improve HIV disease progression.

One of the first-line treatments for trauma in non-HIV populations is Eye Movement Desensitization and Reprocessing (EMDR) therapy. EMDR is a psychotherapeutic approach developed in the late 80s by Francine Shapiro that aims to treat traumatic memories and their associated stress symptoms. This therapy consists of a standard protocol which includes eight phases and bilateral stimulation (usually horizontal saccadic eye movements) to desensitize the discomfort caused by traumatic memories and the aim of the therapy is to achieve their reprocessing and integration within the patient's standard biographical memories. EMDR therapy is recommended by the World Health Organization as a psychotherapy of choice in the treatment of PTSD, showing efficacy in children, teenagers, and adults. Recent studies show potential for EMDR as an efficacious treatment in non-PTSD patients, including in promoting treatment adherence in bipolar patients and as an add-on treatment in chronic pain conditions, as per a recent review. Therefore, EMDR would seem to be indicated as an interesting therapeutic tool in helping people successfully assimilate the HIV diagnosis and reduce psychological distress and psychological trauma symptoms, and as an adjuvant treatment to health-related quality of life and potentially treatment adherence and biological markers of the disease.

This study aims to be the first to test the efficacy of the EMDR therapy in people recently diagnosed with HIV. If shown to be efficacious in this population, it could open the way for future studies to test the efficacy of EMDR in reducing risk behaviors associated with HIV transmission and as a treatment adjunct in treatment-refractory patients.

Evaluation & Diagnostic Protocol

In the baseline visit, sociodemographic data will be taken through a data collection notebook (CRD) and the validated Spanish versions of clinical scales, as well as scales related to health-related quality of life and functionality will be administered. At 6 months, the measures will be taken again, along with a measure regarding satisfaction of the treatment for participants in the EMDR group.

Side Effects and Follow Up

EMDR therapy is a safe and well tolerated psychological treatment. However, some may feel discomfort or suffer when the horizontal eye movements are carried out. If this occurs, bilateral stimulation will be achieved via tapping, which consists of small taps on the hands. Likewise, therapeutic work on difficult life experiences can accentuate psychological distress symptoms. The patient will be taught a variety of self-control techniques to be able to deal with the disturbing information which may arise during and between sessions. Any incident will be registered in the patient's clinical history as well as the CRD of the investigation project to later report the data.

Data Collection: Selection and Evaluation of Study Sample

Study participation is voluntary after being informed of the study objectives and having signed the informed consent document. The participants will be evaluated individually by specially trained health professionals (psychiatrists and psychologists qualified to make diagnoses). The project has been sent and approved to the Ethical Committee for Clinical Investigations in our Centre (number nº 2018/8199/I). Following the baseline evaluation, randomization will be carried out, stratified by age, sex and presence of prior trauma. Data will be collected post intervention. Motives for refusal to participate in the study will be collected to determine the presence of selection bias in the sample and the causes of non-participation.

Statistical Analysis

Calculation of Sample Size:

The study aims to evaluate the efficacy of the EMDR intervention protocol with TAU compared to TAU-only in terms of reduction of posttraumatic symptoms and psychological distress and an improvement in functionality, health-related quality of life, treatment adherence, and the biological markers of HIV of CD4 and the CD4/CD8 ratio. More specifically, the study will evaluate the efficacy of the EMDR therapy compared to treatment as usual in patients with HIV and psychological trauma in terms of clinical stabilization and improvement: reduction of associated trauma and affective symptoms, improvement of functioning, health-related quality of life and biological markers. This is a pilot study in order to get a signal whether or not this intervention is helpful with a planned sample size of 40. However, all patients meeting the inclusion criteria will be assigned to EMDR (n=20) or the TAU group (n=20) by two independent researchers using to the following algorithm: The first two patients will be randomly allocated to EMDR or TAU. For each subsequent patient, the treatment allocation will be identified, which a) balances the arm sizes if one arm has two patients more than the other arm, or otherwise b) decreases the largest effect-size of the between-arms differences in age, sex and trauma type. All steps of the randomization process will be automatically carried out in a central location using a computer program. Effect sizes will be estimated using Hedge's g, directly calculated in numeric variables and converted from odds ratios in binary variables.

Analysis of the main study variables

The distribution of the between-group socio-demographic and clinical characteristics at baseline will be analyzed using descriptive statistics. The continuous variables with a normal distribution will be analyzed with a Multivariate Analysis of Variance (MANOVA). The change in clinical and biological variables compared to baseline at strategic times during the intervention will be analyzed using an ANOVA with repeated measures including time factors, treatment conditions and their interaction. For cases which do not meet the normality premise, the Wilcoxon test will be used. The differences between groups, for the categorical and main clinical variables, will be analyzed using the Chi-squared test. Those variables which are statistically significant can be used as covariables in a logistical regression or lineal study of the factors associated with the significance of the effect, and to determine which variables are the best predictors of function. The effect size index will be estimated (Hedge's g or Pearson's r) for the correlation index of each analysis carried out. The statistical software used for all analyses will be the latest available version of SPSS (v. 24).

Analysis of Clinical Efficacy

For the main statistical analysis, the Intention to Treat (ITT) principal will be applied. The Last Observation Carried Forward (LOCF) will be used as the measure in cases of dropout.

Ethical Issues

The current Project will be carried out in accordance with the basic principles of protection of human rights and dignity as per the Helsinki Declaration and as per current legislation. The study will not begin until the Ethical Committee for Clinical Investigations (CEIC) gives approval and all information gathered will be treated confidentially, as per EU Regulation 2016/679. Patients will be informed verbally and need to sign the attached informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV within last 1 month
* Aged 18 - 65
* Impact of Events Scale-Revised score of higher than 0 related to HIV diagnosis
* Fluency in Spanish
* Initiating antiretroviral medication

Exclusion Criteria:

* Diagnosis of severe mental disorder or neurological disorder
* Current suicidal ideation
* Current substance use disorder
* Have received a structured therapy for trauma in the past 2 years (for part 2 of the study only)
* Clinical diagnosis of AIDS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Psychological trauma | From baseline to posttreatment at 6 months
  Psychological trauma will be evaluated using the Impact of Events Scale-Revised. This scale consists in 22-item to determine frequency and impact of posttraumatic symptoms experienced, with subscales of intrusion, avoidance and hyperarousal, each scored on a 5-point Likert scale, yielding a score for each subscale and a total score. This scale has a scoring range of 0 to 88. On this test, scores that exceed 24 can be quite meaningful. High scores have the following associations: 24 or more PTSD is a clinical concern. Those with scores this high who do not have full PTSD will have partial PTSD or at least some of the symptoms; 33 and above represents the best cutoff for a probable diagnosis of PTSD; 37 or more this is high enough to suppress your immune system's functioning (even 10 years after an impact event).

SECONDARY OUTCOMES:
Post-traumatic stress disorder | From baseline to posttreatment at 6 months
  Post-traumatic stress disorder will be assessed using the Global Post-traumatic Stress Evaluation-DSM V (EGEP-5). This scale consists a 58-item self-report checklist of posttraumatic symptoms to enable diagnosis as per DSM-V criteria. The items are separated in three sections: events (27 items), symptoms (28 items) and functioning (7 items). The scale has been designed to obtain information about: posttraumatic stress disorder (PTSD), intensity or severity of the posttraumatic symptoms (using scales), number of current posttraumatic symptoms, intensity or gravity of the subjective clinical symptoms, disorder specification (chronic or intense PTSD and its beginning), and the level of functional damage.
Dissociative symptoms | From baseline to posttreatment at 6 months
  Dissociation will be evaluated using the Dissociative Experiences Scale (DES). This scale consists a 28-item self-report scale to identify the presence of 3 main symptom clusters of dissociation: amnesia, depersonalization and absorption. Scores are obtained for each subscale from 0 (occurring 0% of times) to 100 (occurring 100% of the time). There is also a global score and can be obtained by summing all the values of the items and dividing them by 28. The higher DES score means the more likely is that the patient has a dissociative disorder.
Anxiety | From baseline to posttreatment at 6 months
  Anxiety will be assessed using the Generalized Anxiety Disorder-7 scale (GAD-7). This scales consists a 7-item self-administered scale to measure the severity of anxiety symptoms over the last 2 weeks and to screen between the anxiety disorders (Generalized Anxiety Disorder, Panic Disorder, Social Phobia and Post Traumatic Stress Disorder). Each item is scored on a 3-point Likert scale, with a cut-off score of 10 indicating clinical symptoms. The global score can be obtained by summing all the answers of the items. Higher scores correlate with disability and functional impairment.
Depression | From baseline to posttreatment at 6 months
  Depression will be evaluated using the Patient Health Questionnaire-9 (PHQ-9). This scale consists a self-administered depression rating scale based on 9 items. Each of the items checked as positive have to be answered in a 3-point Likert scale. The global score can be obtained by summing all the answers of the items. The cut-off score of 10 indicates clinical symptoms (1-4 scores show minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression and 20-27 severe depression).
General psychopathology | From baseline to posttreatment at 6 months
  General psychopathology will be assessed using the Brief Psychiatric Rating Scale (BPRS). This scale is used to assess the gravity and sub-classification (negative or positive) of the schizophrenic disorder. Each item is scored on a 7-point Likert scale, between 1 (symptom absence) and 7 (extremely severe). The total score is obtained summing the scores of each of the 18 items, ranging between 18 and 126. The score of the negative symptoms cluster is obtained by adding the scores of the following items: 3, 13, 16 and 18. This punctuation ranges between 4 and 28. The score of the positive symptoms cluster is obtained by adding the scores of the following items: 4, 11, 12 and 15. This punctuation also ranges between 4 and 28.
Perception of quality of life | From baseline to posttreatment at 6 months
  Quality of life will be evaluated using the Medical Outcomes Study-Short Form 30 items (MOS-HIV 30). This scale consists a 35-item self-report in 11 domains to assess eleven dimensions of health including General Health Perceptions, Pain, Physical Functioning, Role Functioning, Social Functioning, Mental Health, Energy/Fatigue, Health Distress, Cognitive Function, Quality of Life and Health Transition. The raw scores for each scale are transformed to a 0-100 scale, with higher scores indicating a better quality of life and functioning.
Treatment adherence | From baseline to posttreatment at 6 months
  Adherence to pharmacological treatment will be evaluated using the Morisky scale. The Morisky scale is designed to estimate the risk of medication non-adherence. Scores are based on patient responses to four, Yes or No questions. The total scores are ranked from 0 to 4, where the highest scores reflect greater medication adherence.
CD4T and CD8T cells | From baseline to posttreatment at 6 months
  The average levels of CD4T and in the CD4T/CD8T index will be measured using blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt L Amann, PhD, Principal Investigator — Parc de Salut Mar; Fundación IMIM; Universitat Autónoma de Barcelona; CIBERSAM
Locations (1):
- Parc de Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Currently there are no plans.

REFERENCES:
- [Background] Brezing C, Ferrara M, Freudenreich O. The syndemic illness of HIV and trauma: implications for a trauma-informed model of care. Psychosomatics. 2015 Mar-Apr;56(2):107-18. doi: 10.1016/j.psym.2014.10.006. Epub 2014 Oct 8. PMID 25597836
- [Background] Brief DJ, Bollinger AR, Vielhauer MJ, Berger-Greenstein JA, Morgan EE, Brady SM, Buondonno LM, Keane TM; HIV/AIDS Treatment Adherence, Health Outcomes and Cost Study Group. Understanding the interface of HIV, trauma, post-traumatic stress disorder, and substance use and its implications for health outcomes. AIDS Care. 2004;16 Suppl 1:S97-120. doi: 10.1080/09540120412301315259. PMID 15736824
- [Background] Creswell JD, Myers HF, Cole SW, Irwin MR. Mindfulness meditation training effects on CD4+ T lymphocytes in HIV-1 infected adults: a small randomized controlled trial. Brain Behav Immun. 2009 Feb;23(2):184-8. doi: 10.1016/j.bbi.2008.07.004. Epub 2008 Jul 19. PMID 18678242
- [Background] Gonzalez-Garcia M, Ferrer MJ, Borras X, Munoz-Moreno JA, Miranda C, Puig J, Perez-Alvarez N, Soler J, Feliu-Soler A, Clotet B, Fumaz CR. Effectiveness of Mindfulness-Based Cognitive Therapy on the Quality of Life, Emotional Status, and CD4 Cell Count of Patients Aging with HIV Infection. AIDS Behav. 2014 Apr;18(4):676-685. doi: 10.1007/s10461-013-0612-z. Epub 2013 Sep 28. PMID 24077971
- [Background] Gonzalez A, Locicero B, Mahaffey B, Fleming C, Harris J, Vujanovic AA. Internalized HIV Stigma and Mindfulness: Associations With PTSD Symptom Severity in Trauma-Exposed Adults With HIV/AIDS. Behav Modif. 2016 Jan;40(1-2):144-63. doi: 10.1177/0145445515615354. Epub 2015 Nov 19. PMID 26584609
- [Background] Hansen NB, Brown LJ, Tsatkin E, Zelgowski B, Nightingale V. Dissociative experiences during sexual behavior among a sample of adults living with HIV infection and a history of childhood sexual abuse. J Trauma Dissociation. 2012;13(3):345-60. doi: 10.1080/15299732.2011.641710. PMID 22545567
- [Background] Jam S, Imani AH, Foroughi M, SeyedAlinaghi S, Koochak HE, Mohraz M. The effects of mindfulness-based stress reduction (MBSR) program in Iranian HIV/AIDS patients: a pilot study. Acta Med Iran. 2010 Mar-Apr;48(2):101-6. PMID 21133002
- [Background] Jonas DE, Cusack K, Forneris CA, Wilkins TM, Sonis J, Middleton JC, Feltner C, Meredith D, Cavanaugh J, Brownley KA, Olmsted KR, Greenblatt A, Weil A, Gaynes BN. Psychological and Pharmacological Treatments for Adults With Posttraumatic Stress Disorder (PTSD) [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Apr. Report No.: 13-EHC011-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK137702/ PMID 23658937
- [Background] Siyahhan Julnes P, Auh S, Krakora R, Withers K, Nora D, Matthews L, Steinbach S, Snow J, Smith B, Nath A, Morse C, Kapetanovic S. The Association Between Post-traumatic Stress Disorder and Markers of Inflammation and Immune Activation in HIV-Infected Individuals With Controlled Viremia. Psychosomatics. 2016 Jul-Aug;57(4):423-30. doi: 10.1016/j.psym.2016.02.015. Epub 2016 Mar 2. PMID 27095586
- [Background] Katz S, Nevid JS. Risk factors associated with posttraumatic stress disorder symptomatology in HIV-infected women. AIDS Patient Care STDS. 2005 Feb;19(2):110-20. doi: 10.1089/apc.2005.19.110. PMID 15716642
- [Background] Knobel H, Carmona A, Grau S, Pedro-Botet J, Diez A. Adherence and effectiveness of highly active antiretroviral therapy. Arch Intern Med. 1998 Sep 28;158(17):1953. doi: 10.1001/archinte.158.17.1953. No abstract available. PMID 9759698
- [Background] Machtinger EL, Wilson TC, Haberer JE, Weiss DS. Psychological trauma and PTSD in HIV-positive women: a meta-analysis. AIDS Behav. 2012 Nov;16(8):2091-100. doi: 10.1007/s10461-011-0127-4. PMID 22249954
- [Background] McEwen BS, Seeman T. Protective and damaging effects of mediators of stress. Elaborating and testing the concepts of allostasis and allostatic load. Ann N Y Acad Sci. 1999;896:30-47. doi: 10.1111/j.1749-6632.1999.tb08103.x. PMID 10681886
- [Background] Moreno-Alcazar A, Treen D, Valiente-Gomez A, Sio-Eroles A, Perez V, Amann BL, Radua J. Efficacy of Eye Movement Desensitization and Reprocessing in Children and Adolescent with Post-traumatic Stress Disorder: A Meta-Analysis of Randomized Controlled Trials. Front Psychol. 2017 Oct 10;8:1750. doi: 10.3389/fpsyg.2017.01750. eCollection 2017. PMID 29066991
- [Background] Mugavero M, Ostermann J, Whetten K, Leserman J, Swartz M, Stangl D, Thielman N. Barriers to antiretroviral adherence: the importance of depression, abuse, and other traumatic events. AIDS Patient Care STDS. 2006 Jun;20(6):418-28. doi: 10.1089/apc.2006.20.418. PMID 16789855
- [Background] Mugavero MJ, Raper JL, Reif S, Whetten K, Leserman J, Thielman NM, Pence BW. Overload: impact of incident stressful events on antiretroviral medication adherence and virologic failure in a longitudinal, multisite human immunodeficiency virus cohort study. Psychosom Med. 2009 Nov;71(9):920-6. doi: 10.1097/PSY.0b013e3181bfe8d2. Epub 2009 Oct 29. PMID 19875634
- [Background] Nightingale VR, Sher TG, Mattson M, Thilges S, Hansen NB. The effects of traumatic stressors and HIV-related trauma symptoms on health and health related quality of life. AIDS Behav. 2011 Nov;15(8):1870-8. doi: 10.1007/s10461-011-9980-4. PMID 21667297
- [Background] Nightingale VR, Sher TG, Hansen NB. The impact of receiving an HIV diagnosis and cognitive processing on psychological distress and posttraumatic growth. J Trauma Stress. 2010 Aug;23(4):452-60. doi: 10.1002/jts.20554. PMID 20648562
- [Background] Novo P, Landin-Romero R, Radua J, Vicens V, Fernandez I, Garcia F, Pomarol-Clotet E, McKenna PJ, Shapiro F, Amann BL. Eye movement desensitization and reprocessing therapy in subsyndromal bipolar patients with a history of traumatic events: a randomized, controlled pilot-study. Psychiatry Res. 2014 Sep 30;219(1):122-8. doi: 10.1016/j.psychres.2014.05.012. Epub 2014 May 15. PMID 24880581
- [Background] Pence BW, Mugavero MJ, Carter TJ, Leserman J, Thielman NM, Raper JL, Proeschold-Bell RJ, Reif S, Whetten K. Childhood trauma and health outcomes in HIV-infected patients: an exploration of causal pathways. J Acquir Immune Defic Syndr. 2012 Apr 1;59(4):409-16. doi: 10.1097/QAI.0b013e31824150bb. PMID 22107822
- [Background] Seedat S, Stein DJ, Carey PD. Post-traumatic stress disorder in women: epidemiological and treatment issues. CNS Drugs. 2005;19(5):411-27. doi: 10.2165/00023210-200519050-00004. PMID 15907152
- [Background] SeyedAlinaghi S, Jam S, Foroughi M, Imani A, Mohraz M, Djavid GE, Black DS. Randomized controlled trial of mindfulness-based stress reduction delivered to human immunodeficiency virus-positive patients in Iran: effects on CD4(+) T lymphocyte count and medical and psychological symptoms. Psychosom Med. 2012 Jul-Aug;74(6):620-7. doi: 10.1097/PSY.0b013e31825abfaa. Epub 2012 Jun 28. PMID 22753635
- [Background] Shapiro F. Eye movement desensitization: a new treatment for post-traumatic stress disorder. J Behav Ther Exp Psychiatry. 1989 Sep;20(3):211-7. doi: 10.1016/0005-7916(89)90025-6. PMID 2576656
- [Background] Sherr L, Nagra N, Kulubya G, Catalan J, Clucas C, Harding R. HIV infection associated post-traumatic stress disorder and post-traumatic growth--a systematic review. Psychol Health Med. 2011 Oct;16(5):612-29. doi: 10.1080/13548506.2011.579991. Epub 2011 Jul 27. PMID 21793667
- [Background] Theuninck AC, Lake N, Gibson S. HIV-related posttraumatic stress disorder: investigating the traumatic events. AIDS Patient Care STDS. 2010 Aug;24(8):485-91. doi: 10.1089/apc.2009.0231. PMID 20632886
- [Background] Valiente-Gomez A, Moreno-Alcazar A, Treen D, Cedron C, Colom F, Perez V, Amann BL. EMDR beyond PTSD: A Systematic Literature Review. Front Psychol. 2017 Sep 26;8:1668. doi: 10.3389/fpsyg.2017.01668. eCollection 2017. PMID 29018388
- [Background] Vranceanu AM, Safren SA, Lu M, Coady WM, Skolnik PR, Rogers WH, Wilson IB. The relationship of post-traumatic stress disorder and depression to antiretroviral medication adherence in persons with HIV. AIDS Patient Care STDS. 2008 Apr;22(4):313-21. doi: 10.1089/apc.2007.0069. PMID 18338960
- [Background] Young C. Understanding HIV-related posttraumatic stress disorder in South Africa: a review and conceptual framework. Afr J AIDS Res. 2011 Jun;10(2):139-48. doi: 10.2989/16085906.2011.593376. PMID 25859736
- [Background] Guidelines for the Management of Conditions Specifically Related to Stress. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK159725/ PMID 24049868
- [Background] Hase, M. (2018). Medical Trauma: EMDR Therapy to Treat the Sequelae of Somatic Illness and Medical Treatment. In M. Luber (Ed.), Eye Movement Desensitization and Reprocessing (EMDR) Therapy Scripted Protocols and Summary Sheets: Treating Trauma in Somatic and Medical Related Conditions. New York: Springer Publishing Company.
- [Background] Shapiro, F. (2005). Desensibilización y Reprocesamiento Por Movimiento Ocular (2nd ed.). México: Pax.